CLINICAL TRIAL: NCT04185636
Title: Prospective, Double-blind Assessment of the Presence of Fluorescence Signature to Predict Graft Failure Using MolecuLight i:X Imaging Device
Brief Title: Presence of Fluorescence Signature to Predict Graft Failure Using MolecuLight i:X
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-003
Record Dates: First submitted 2019-11-29; First posted 2019-12-04 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Skin Graft (Allograft)(Autograft) Failure
Keywords: Bacterial fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Skin Graft Patients: There will only be 1 group, patients receiving a skin graft and MolecuLight i:X imaging
  Interventions: Device: MolecuLight i:X imaging

INTERVENTIONS:
Device: MolecuLight i:X imaging — The MolecuLight i:X Imaging Device will be used to take standard (ST) and fluorescent (FL) images of each graft site. The MolecuLight i:X will also be used to take measurements of the wound using the measurement feature of the device.

SUMMARY:
This study will investigate whether the presence of a bacterial fluorescent signature captured by the MolecuLight i:X can predict a skin graft failure. The MolecuLight i:X is a handheld medical device which enables real-time standard digital imaging and fluorescence imaging of wounds and surrounding healthy skin of patients. When wounds are illuminated in fluorescence mode, collagen and other related proteins in the connective tissue matrix may emit a characteristic green fluorescent signal, while some bacteria may emit a unique red fluorescence signal due to endogenous porphyrin production and others may emit a unique cyan fluorescence signal due to the production of pyoverdine.

This is a non-randomized evaluation for which 20 adult patients will be imaged at University Hospitals Birmingham who present with a wound which has been previously infected and which requires a skin graft. The i:X will be used to take standard and fluorescent (FL) images of each graft site by the study team. The wound will be measured using the measurement application of the i:X, using WoundStickers. The clinician will be blinded to the results of these FL images until the end of the study. In this trial, the device is not intended to guide treatment. The images will be used after a 1-month patient follow up to correlate presence of bacterial fluorescence signature to graft failure. The hypothesis is that the presence of a bacterial fluorescence signature increases the likelihood of graft failure. The ability to predict graft failure would provide clinicians with more information on which to base a patient's suitability for a graft (e.g. determining if there is a heavy bacterial load present). This may lead to selection of appropriate therapies before a graft is applied.

DETAILED DESCRIPTION:
This is a non-randomized evaluation for which 20 adult patients will be imaged at University Hospitals Birmingham who present with a wound which has been previously infected and which requires a skin graft. The MolecuLight i:X Imaging Device will be used to take standard (ST) and fluorescent (FL) images of each graft site. The MolecuLight i:X will also be used to take measurements of the wound using the measurement feature of the device.

Once a patient has identified as being suitable for the trial, the study will be introduced to them by a member of their circle of care. They will be provided with an informed consent form, provided time to consider the study and have any of their questions answered. The patient will be asked to sign and date the ICF if they choose to participate in the study.The subjects will be recruited for a period of 2 months.

The execution of the full protocol is expected to take approximately 15 minutes during a single clinic visit for each study subject. During the clinic visit, the clinician will treat the patient based on their clinical practice. Prior to the application of the skin graft, the Moleculight i:X will be used to take standard and fluorescent (FL) images of each graft site by the study team. The wound will be measured using the measurement application of the i:X, using WoundStickers. Following imaging the skin graft will be applied and treatment will continue as per the clinician's clinical practice.

The clinician will be blinded to the results of these FL images until the end of the study. In this trial, the device is not intended to guide treatment. There will be a follow-up with each patient at 1 month after the grafting procedure to ask if the grafting procedure was successful. There will not be any imaging or sampling required at the time of follow-up. The information gathered will be used for post-hoc analysis to assess if the presence of a fluorescence signal at the time of imaging is correlated to graft failure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a wound with previous infection, requiring a skin graft
* 18 years or older

Exclusion Criteria:

* Subject has been treated with an investigational drug within 1 month before enrollment
* Subject is unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at 1 clinical site in the United Kingdom with a wound with a previous infection requiring a skin graft.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Graft success or failure | 1 month
  Correlation between presence of bacterial fluorescence signature in a wound and failure of a graft.

SECONDARY OUTCOMES:
Economic Analysis | 1 month
  Estimate the cost benefit of identifying and resolving an infection prior to graft (a. Estimate cost of graft procedure without complications, b. Estimate health care and quality of life cost of graft that becomes infected (initial graft, resolution of infection, secondary graft procedures, etc.), c. Estimate health care and quality of life cost of identifying infection prior to initial graft, resolve infection, and then graft procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jeffery, MB ChB, Principal Investigator — Birmingham City University Hospitals
Locations (1):
- Birmingham City University Hospitals, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study will not make IPD available to other researchers.